CLINICAL TRIAL: NCT02322814
Title: A Multistage, Phase II Study Evaluating the Safety and Efficacy of Cobimetinib Plus Paclitaxel, Cobimetinib Plus Atezolizumab Plus Paclitaxel, or Cobimetinib Plus Atezolizumab Plus Nab-Paclitaxel as First-Line Treatment for Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Cobimetinib Plus Paclitaxel, Cobimetinib Plus Atezolizumab Plus Paclitaxel, or Cobimetinib Plus Atezolizumab Plus Nab-Paclitaxel as Initial Treatment for Participants With Triple-Negative Breast Cancer That Has Spread
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29479; 2014-002230-32 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — cobimetinib; Paclitaxel; atezolizumab; 130-nm albumin-bound paclitaxel

ARMS (4):
- Cohort I: Cobimetinib, Paclitaxel (Experimental): Participants will receive a combination of cobimetinib plus paclitaxel in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
  Interventions: Drug: Cobimetinib; Drug: Paclitaxel
- Cohort I: Placebo, Paclitaxel (Placebo Comparator): Participants will receive a combination of cobimetinib placebo plus paclitaxel in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
  Interventions: Drug: Paclitaxel; Drug: Placebo
- Cohort II:Cobimetinib,Paclitaxel,Atezolizumab (Experimental): Participants will receive cobimetinib plus paclitaxel plus atezolizumab in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
  Interventions: Drug: Cobimetinib; Drug: Paclitaxel; Drug: Atezolizumab
- Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab (Experimental): Participants will receive cobimetinib plus nab-paclitaxel plus atezolizumab until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be administered orally at a dose of 60 milligrams (mg) per day, once a day, on Day 3 through Day 23 of each 28-day treatment cycle.
  Other Names: GDC-0973; RO5514041; XL518
  Arms: Cohort I: Cobimetinib, Paclitaxel; Cohort II:Cobimetinib,Paclitaxel,Atezolizumab; Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 80 milligrams per square meter (mg/m^2) by intravenous (IV) infusion on Day 1, Day 8, and Day 15 of each 28-day cycle according to prescribing information.
  Arms: Cohort I: Cobimetinib, Paclitaxel; Cohort I: Placebo, Paclitaxel; Cohort II:Cobimetinib,Paclitaxel,Atezolizumab
Drug: Placebo — Placebo matching to cobimetinib will be administered orally, once a day, on Day 3 through Day 23 of each 28 day treatment cycle.
  Arms: Cohort I: Placebo, Paclitaxel
Drug: Atezolizumab — Atezolizumab will be administered to Cohorts II and III at a dose of 840 mg IV every 2 weeks on Days 1 and 15 of each 28-day treatment cycle.
  Other Names: MPDL3280A
  Arms: Cohort II:Cobimetinib,Paclitaxel,Atezolizumab; Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered to Cohort III according to the local prescribing information at a starting dose of 100 mg/m^2 by IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Arms: Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab

SUMMARY:
This three-cohort, multi-stage, randomized, Phase II, multicenter trial will evaluate the safety and tolerability and estimate the efficacy of cobimetinib plus paclitaxel versus placebo plus paclitaxel in Cohort I, of cobimetinib plus atezolizumab plus paclitaxel in Cohort II, and of cobimetinib plus atezolizumab plus nab-paclitaxel in Cohort III in participants with metastatic or locally advanced, triple-negative adenocarcinoma of the breast who have not received prior systemic therapy for metastatic breast cancer (MBC). Participants may continue on study treatment until the development of progressive disease (PD) or the loss of clinical benefit, unacceptable toxicity, and/or consent withdrawal. The Cohort I target sample size is 12 participants for the safety run-in stage and approximately 90 participants in the expansion stage. Each of Cohorts II and III will consist of a safety run-in stage of approximately 15 participants followed by an expansion stage of approximately 15 participants.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and human epidermal growth factor 2 (HER2)-negative adenocarcinoma of the breast with measurable metastatic or locally advanced disease
* Locally advanced disease must not be amenable to resection with curative intent
* Measurable disease, according to RECIST, v1.1
* Adequate hematologic and end organ function
* Agreement to use highly effective contraceptive methods as stated in protocol

Exclusion Criteria:

Disease-Specific Exclusion Criteria

* Known HER2-, ER-positive, or PR-positive breast cancer by local laboratory assessment
* Any prior chemotherapy, hormonal, or targeted therapy, for inoperable locally advanced or metastatic triple-negative breast cancer (mTNBC)
* Any systemic anticancer therapy within 3 weeks prior to Cycle 1, Day 1
* Any radiation treatment to metastatic site within 28 days of Cycle 1, Day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Cycle 1, Day 1 or anticipation of need for major surgical procedure during the course of the study
* Prior exposure to experimental treatment targeting rapidly accelerated fibrosarcoma (Raf), MAP kinase/ERK kinase (MEK), or the mitogen-activated protein kinase (MAPK) pathway
* Brain metastases (symptomatic or nonsymptomatic) that have not been treated previously, are progressive, or require any type of therapy (e.g., radiation, surgery, or steroids) to control symptoms from brain metastases within 30 days prior to first study treatment dose

Cobimetinib-Specific Exclusion Criteria

* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* Cobimetinib is metabolized by the hepatic cytochrome P3A4 (CYP3A4) enzyme. Drugs CYP3A4/5 inhibitors and inducers should be avoided

Atezolizumab-Specific Exclusion Criteria (Cohorts II and III Only)

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease
* Prior allogenic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive test for Human Immunodeficiency Virus (HIV)
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] or positive hepatitis B virus [HBV] deoxyribonucleic acid [DNA] test at screening) or hepatitis C
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to randomization or anticipation that such a live, attenuated vaccine will be required during the study
* Prior treatment with cluster of differentiation (CD) 137 (CD137) agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), or anti-programmed death ligand-1 (anti-PD-L1) therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or Interlukin-2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial

Cardiac Exclusion Criteria

* History of clinically significant cardiac dysfunction
* Corrected QT interval at screening greater than (>) 480 milliseconds (ms) (average of triplicate screening measurements)
* Left ventricular ejection fraction (LVEF) below the institutional lower limit of normal or below 50 percent (%), whichever is lower

General Exclusion Criteria

* No other history of or ongoing malignancy that would potentially interfere with the interpretation of the pharmacodynamic or efficacy assay
* Pregnancy (positive serum pregnancy test) or lactation
* Uncontrolled serious medical or psychiatric illness
* Active infection requiring IV antibiotics on Cycle 1, Day 1
* Participants who have a history of hypersensitivity reactions to paclitaxel or other drugs formulated in Cremophor® EL (polyoxyethylated castor oil) or to nab-paclitaxel and any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (11):
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mercy Hospital, a Campus of Plantation General Hospital, Miami, Florida
  - Florida Hospital Cancer Inst, Orlando, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (4):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - St John of God Murdoch Hospital; Oncology West, Murdoch, Western Australia
- Belgium (5):
  - Clinique Edith Cavell, Brussels
  - AZ Sint Lucas (Sint Lucas), Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - AZ Sint Augustinus Veurne, Veurne
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Multiscan s.r.o., Pardubice
- France (4):
  - Centre Oscar Lambret, Lille
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - Hopital Tenon, Paris
  - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer, Rennes
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (6):
  - Azienda Ospedaliero Universitaria Seconda Università Degli Studi Di Napoli, Napoli, Campania
  - A.O.U Policlinico S. Orsola Malpighi di Bologna U.O di Medicina Interna Borghi - Pad.2, Bologna, Emilia-Romagna
  - Centro Di Riferimento Oncologico; SOC Oncologia Medica C, Aviano, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Ospedaliero - Universitaria Pisana U.O. Oncologia Medica 2 Universitaria ? Polo Oncologico, Pisa, Tuscany
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- Romania (2):
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
- South Korea (4):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
- Spain (7):
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Organización Sanitaria Integrada Bilbao Basurto, Bilbao, Vizcaya
  - Hospital Universitario Infanta Cristina; Servicio de Oncologia, Badajoz
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Nefrologia, Madrid
  - Hosp. Regional Univ. de Malaga ? Hospital Materno Infantil; Hospital Materno Infantil de Malaga, Málaga
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung Country
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
- United Kingdom (3):
  - Nuffield Health Bournemouth Hospital, Bournemouth
  - Mount Vernon Hospital, Middlesex
  - Nottingham University Hospitals City Campus, Nottingham

REFERENCES:
- [Derived] Barteselli G, Goodman GR, Patel Y, Caro I, Xue C, McCallum S. Characterization of Serous Retinopathy Associated with Cobimetinib: Integrated Safety Analysis of Four Studies. Drug Saf. 2022 Dec;45(12):1491-1499. doi: 10.1007/s40264-022-01248-2. Epub 2022 Oct 30. PMID 36310331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants with metastatic or locally advanced, triple-negative adenocarcinoma of the breast who had not received prior systemic therapy for metastatic breast cancer. Locally advanced disease must not have been amenable to resection with curative intent.
Pre-assignment Details: One participant from Cohort III never started any treatment.
Groups:
- Cohort I: Safety Run-In: Participants received cobimetinib plus paclitaxel until 12 participants completed one cycle of study treatment (28 days).
- Cohort I: Placebo, Paclitaxel: Participants received a combination of cobimetinib placebo plus paclitaxel in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
- Cohort I: Cobimetinib, Paclitaxel: Participants received a combination of cobimetinib plus paclitaxel in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
- Cohort II:Cobimetinib,Paclitaxel,Atezolizumab: Participants received cobimetinib plus paclitaxel plus atezolizumab in 28-day cycles until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
- Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab: Participants received cobimetinib plus nab-paclitaxel plus atezolizumab until disease progression, unacceptable toxicity, investigator decision, death, withdrawal of consent, or completion of study.
Period: Overall Study
Arm/Group | Cohort I: Safety Run-In | Cohort I: Placebo, Paclitaxel | Cohort I: Cobimetinib, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Started | 16 | 43 | 47 | 32 | 31
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 43 | 47 | 32 | 31
Not completed — Death | 7 | 29 | 32 | 23 | 14
Not completed — Lost to Follow-up | 1 | 3 | 3 | 1 | 0
Not completed — Various Reasons | 2 | 0 | 1 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 7 | 9 | 5 | 13
Not completed — Withdrawal by Subject | 5 | 4 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all enrolled participants, whether or not the assigned study treatment was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: Safety Run-In | Cohort I: Placebo, Paclitaxel | Cohort I: Cobimetinib, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab | Total
Number analyzed (Participants) | 16 | 43 | 47 | 32 | 31 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (12.7) | 52.9 (13.7) | 54.2 (10.3) | 53.7 (13.1) | 52.2 (11.8) | 53.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 43 | 47 | 32 | 31 | 169
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 3 | 2 | 3 | 16
  Not Hispanic or Latino | 13 | 35 | 41 | 30 | 28 | 147
  Unknown or Not Reported | 2 | 1 | 3 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 9 | 11 | 2 | 5 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 1 | 0 | 5
  White | 10 | 34 | 32 | 28 | 25 | 129
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cohort I: Progression-Free Survival, as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression or relapse, as determined by the investigator, using RECIST v1.1. As per RECIST v1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: Randomization up to disease progression or relapse, whichever occurs first (up to approximately 2 years)
Population: ITT population was defined as all enrolled participants, whether or not the assigned study treatment was received. Data were only collected from participants in the Cohort I Expansion Stage (Cohort I: Cobimetinib, Paclitaxel, Cohort I: Placebo, Paclitaxel) for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel
Number analyzed (Participants) | 47 | 43
Weeks | 23.71 [18.14 to 32.14] | 16.43 [8.14 to 31.14]
Statistical Analysis 1: Comparison: Cohort I: Cobimetinib, Paclitaxel vs Cohort I: Placebo, Paclitaxel; Test type: Superiority; p = 0.2470, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI [0.43 to 1.24]

2. Primary Outcome: Cohort II, III: Percentage of Participants With Confirmed Overall Response (OR) (Partial Response [PR] or Complete Response [CR]), as Determined by the Investigator Using RECIST v1.1
Description: OR was defined as the rate of a PR or CR occurring after randomization and confirmed >=28 days later as determined by the investigator using RECIST v1.1. As per RECIST v1.1, CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target and new measurable lesions.
Time Frame: Randomization up to disease progression or relapse, whichever occurs first (up to approximately 5.25 years)
Population: ITT population was defined as all enrolled participants, whether or not the assigned study treatment was received.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 32 | 31
Percentage of participants
  Responders | 37.5 | 32.3
  Non-Responders | 62.5 | 67.7

3. Secondary Outcome: Cohort I, II, III: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause
Time Frame: Randomization up to death from any cause (up to approximately 6.5 years)
Population: ITT population was defined as all enrolled participants, whether or not the assigned study treatment was received. Data were only collected from participants in the Cohort I Expansion Stage (Cohort I: Cobimetinib, Paclitaxel, Cohort I: Placebo, Paclitaxel) along with the Cohort II and III for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 47 | 43 | 32 | 31
Months | 16.72 [13.50 to 20.24] | 19.58 [14.75 to 29.37] | 11.04 [9.53 to 22.51] | 15.57 [14.26 to NA] — The upper limit of 95% CI was not evaluable due to insufficient events observed.
Statistical Analysis 1: Comparison: Cohort I: Cobimetinib, Paclitaxel vs Cohort I: Placebo, Paclitaxel; Test type: Superiority; p = 0.5912, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI [0.65 to 2.13]

4. Secondary Outcome: Cohort I: Percentage of Participants With Confirmed OR (PR or CR), as Determined by the Investigator Using RECIST v1.1
Description: as for outcome 2
Time Frame: Randomization up to disease progression or relapse, whichever occurs first (up to approximately 2 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel
Number analyzed (Participants) | 47 | 43
Percentage of participants
  Responders | 38.3 | 20.9
  Non-responders | 61.7 | 79.1

5. Secondary Outcome: Cohort I, II, III: Duration of Response (DOR), as Determined by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the first occurrence of a documented objective response to the time of relapse, as determined by the investigator using RECIST v1.1 or death from any cause during the study, whichever occurred first.
Time Frame: Time from the first occurrence of documented objective response to time of relapse or death, whichever occurs first (up to approximately 6.5 years)
Population: ITT population was defined as all enrolled participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort I: Safety Run-In | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 16 | 47 | 43 | 32 | 31
Months | 39.29 [23.14 to 56.29] | 23.14 [16.14 to 26.57] | 24.14 [17.14 to NA] — The upper limit of 95% CI was not evaluable due to insufficient events observed. | 5.78 [4.44 to 16.33] | 11.42 [5.78 to 17.94]

6. Secondary Outcome: Cohort I, II, III: Percentage of Participants With Unconfirmed Overall Response (OR_uc) (Unconfirmed PR or CR), as Determined by the Investigator Using RECIST v1.1
Description: ORR_uc (ORR confirmation not required) was defined as the rate of a PR or CR occurring after randomization as determined by the investigator using RECIST v1.1, confirmation not required. As per RECIST v1.1, CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target and new measurable lesions.
Time Frame: Randomization up to disease progression or relapse, whichever occurs fist (up to approximately 6.5 years)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 47 | 43 | 32 | 31
Percentage of participants
  Responders | 42.6 | 25.6 | 46.9 | 45.2
  Non-Responders | 57.4 | 74.4 | 53.1 | 54.8

7. Secondary Outcome: Cohort II, III: Progression-Free Survival, as Determined by Investigator Using RECIST v1.1
Description: PFS was defined as the time from randomization to the first occurrence of disease progression or relapse, as determined by the investigator, using RECIST v1.1. As per RECIST v1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Randomization up to disease progression or relapse, whichever occurs first (up to approximately 6.5 years)
Population: ITT population was defined as all enrolled participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 32 | 31
Months | 3.75 [3.02 to 7.29] | 7.66 [3.65 to 11.04]

8. Secondary Outcome: Cohort I, II, III: Percentage of Participants With Adverse Events (AEs)
Time Frame: Randomization up to end of study (up to approximately 6.5 years)
Population: Safety-evaluable population was defined as participants who received any amount of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Safety Run-In | Cohort I: Cobimetinib, Paclitaxel | Cohort I: Placebo, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 16 | 47 | 43 | 32 | 30
Participants | 15 | 46 | 43 | 32 | 30

9. Secondary Outcome: Cohort I, II, III: Maximum Plasma Concentration (Cmax) of Cobimetinib
Time Frame: Safety Run-In: Predose (Hour [Hr] 0) on Cycle (Cy) 1 Day (D) 8; predose (Hr 0), 0.5, 1, 2, 4, 6 Hr postdose (2, 4 Hr postdose for Cohorts II, III) on Cy1 D15; Expansion: predose (Hr 0), 1-4 Hr postdose on Cy1 D15; predose (Hr 0) on Cy2 D15 (Cy=28 days)
Population: The pharmacokinetic (PK) population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilitre (ng/mL)
Arm/Group | Cohort I: Safety Run-In | Cohort I: Cobimetinib, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 11 | 8 | 17 | 15
Nanograms per millilitre (ng/mL) | 285 (62.2) | 266 (82.0) | 213 (68.0) | 407 (90.7)

10. Secondary Outcome: Cohort I, II, III: Minimum Plasma Concentration (Cmin) of Cobimetinib
Time Frame: Safety Run-In: Predose (Hr 0) on Cy 1 D8; predose (Hr 0), 0.5, 1, 2, 4, 6 Hr postdose (2, 4 Hr postdose for Cohorts II, III) on Cy1 D15; Expansion: predose (Hr 0), 1-4 Hr postdose on Cy1 D15; predose (Hr 0) on Cy2 D15 (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Safety Run-In | Cohort I: Cobimetinib, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 13 | 38 | 14 | 13
ng/mL | 65.6 (1279.5) | 130 (190.7) | 138 (79.0) | 136 (67.2)

11. Secondary Outcome: Cohort I: Area Under the Concentration-Time Curve From Time Zero to Dosing Interval (AUC0-tau; Total Exposure) of Cobimetinib
Time Frame: Safety Run-In: Predose (Hr 0) on Cy 1 D8; predose (Hr 0), 0.5, 1, 2, 4, 6 Hr postdose on Cy1 D15; Expansion: predose (Hr 0), 1-4 Hr postdose on Cy1 D15 (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug. Data were only collected from participants in the Cohort I: Safety Run-In stage for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter/hour (hr*ng/mL)
Arm/Group | Cohort I: Safety Run-In
Number analyzed (Participants) | 11
Nanograms/milliliter/hour (hr*ng/mL) | 1620 (80.0)

12. Secondary Outcome: Cohort I, II: Cmax of Paclitaxel
Time Frame: Safety Run-In: Predose (Hr 0) on Cy1 D8; predose (Hr 0), 0.5, 1, 2, 4, and 6 Hr postdose (2, 4 Hr postdose for Cohort II) (infusion duration: 1 Hr) on Cy1 D15 (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug. Data were only collected from Cohort I: Safety Run-In and Cohort II participants for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Safety Run-In | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab
Number analyzed (Participants) | 11 | 14
ng/mL | 1770 (553.4) | 283 (490.9)

13. Secondary Outcome: Cohort I, II: Cmin of Paclitaxel
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Safety Run-In | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab
Number analyzed (Participants) | 13 | 15
ng/mL | 1.40 (89.9) | 1.26 (53.3)

14. Secondary Outcome: Cohort I: AUC0-tau of Paclitaxel
Time Frame: Safety Run-In: Predose (Hr 0) on Cy1 D8; predose (Hr 0), 0.5, 1, 2, 4, and 6 Hr postdose (infusion duration: 1 Hr) on Cy1 D15 (Cy=28 days)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort I: Safety Run-In
Number analyzed (Participants) | 10
hr*ng/mL | 4220 (310.4)

15. Secondary Outcome: Cohort III: Cmax of Nab-Paclitaxel
Time Frame: Safety Run-In: Predose (Hr 0) on Cy1 D8; predose (Hr 0), 2, 4 Hr postdose (infusion duration: 30 minutes) on Cy1 D15 (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 13
ng/mL | 277 (658.5)

16. Secondary Outcome: Cohort III: Cmin of Nab-Paclitaxel
Time Frame: as for outcome 15
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 12
ng/mL | 2.05 (173.9)

17. Secondary Outcome: Cohort III: AUC0-tau of Nab-Paclitaxel
Time Frame: as for outcome 15
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug. Due to the sparse nature of PK sampling, the estimation of this PK parameter requires the use of population PK analysis. This would have enabled the exposure-response analysis with this OM. Given the outcome of the study, the Sponsors did not proceed with popPK analysis, which was planned, only if data warranted. AUC0-tau was not estimated and analyzed using the sparse PK samples.
Arm/Group | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Cohort II, III: Cmax (in Serum) of Atezolizumab
Time Frame: Safety Run-In, Expansion:Predose (Hr0), 0.5Hr postdose (infusion duration:1Hr) on D1 of Cy1, 3; predose (Hr0) on D1 of Cy2, 4, 8, every 8 Cy up to end of treatment (EOT); 120 days after EOT (approximately 5.25 years) (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 10 | 10
ng/mL | 346 (48.3) | 374 (38.8)

19. Secondary Outcome: Cohort II, III: Cmin (in Serum) of Atezolizumab
Time Frame: Safety Run-In, Expansion: Predose (Hr 0), 0.5 Hr postdose (infusion duration: 1 Hr) on D1 of Cy1, 3; predose (Hr 0) on D1 of Cy2, 4, 8, every 8 Cy up to EOT; 120 days after EOT (approximately 5.5 years) (Cy=28 days)
Population: The PK population included all participants with evaluable PK data who received at least one dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 10 | 10
ng/mL | 144 (34.6) | 109 (89.9)

20. Secondary Outcome: Cohort II, III: AUC0-tau (in Serum) of Atezolizumab
Time Frame: Safety Run-In, Expansion: Predose (Hr 0), 0.5 Hr postdose (infusion duration: 1 Hr) on D1 of Cy1, 3; predose (Hr 0) on D1 of Cy2, 4, 8, every 8 Cy up to EOT (approximately 5.5 years); 120 days after EOT (approximately 5.5 years) (Cy=28 days)
Population: as for outcome 17
Arm/Group | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization up until 6.5 years
Description: The All-Cause Mortality table displays information from the ITT population which included all enrolled participants, whether or not the assigned study treatment was received. One participant in Cohort III didn't receive study treatment and is not counted in the AE tables. The safety-evaluable population was defined as participants who received any amount of any study drug. The Serious and Other Adverse Events are reported with data from the safety-evaluable population.
Arm/Group | Cohort I: Safety Run-In | Cohort I: Placebo, Paclitaxel | Cohort I: Cobimetinib, Paclitaxel | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab
All-Cause Mortality (participants affected / at risk) | 7/16 | 29/43 | 32/47 | 23/32 | 14/31
Serious Adverse Events (participants affected / at risk) | 6/16 | 8/43 | 17/47 | 16/32 | 15/30
Other Adverse Events (participants affected / at risk) | 15/16 | 43/43 | 46/47 | 32/32 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I: Safety Run-In (N=16) | Cohort I: Placebo, Paclitaxel (N=43) | Cohort I: Cobimetinib, Paclitaxel (N=47) | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab (N=32) | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab (N=30)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPILLOEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0) | 6 (6) | 4 (4) | 2 (3)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MASTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 2 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMBOLISM VENOUS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I: Safety Run-In (N=16) | Cohort I: Placebo, Paclitaxel (N=43) | Cohort I: Cobimetinib, Paclitaxel (N=47) | Cohort II:Cobimetinib,Paclitaxel,Atezolizumab (N=32) | Cohort III: Cobimetinib, Nab-Paclitaxel, Atezolizumab (N=30)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 6 (9) | 12 (16) | 14 (19) | 10 (24)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (6) | 1 (2) | 1 (1) | 0 (0) | 3 (9)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (16) | 13 (43) | 8 (21) | 6 (6) | 8 (18)
PALPITATIONS (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
CATARACT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT CORTICAL (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 3 (3)
EPISCLERITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
EYELID OEDEMA (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
MACULAR FIBROSIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DRUSEN (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 10 (11) | 4 (4) | 4 (5)
VITREOUS FLOATERS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (6) | 6 (8) | 5 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 4 (5) | 6 (6) | 2 (2) | 1 (1)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 9 (11) | 8 (11) | 6 (7) | 8 (13)
DIARRHOEA (Gastrointestinal disorders) | 10 (29) | 13 (19) | 36 (66) | 21 (48) | 27 (55)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (9) | 1 (1) | 5 (7)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 7 (7) | 18 (25) | 20 (24) | 13 (18) | 15 (20)
STOMATITIS (Gastrointestinal disorders) | 5 (8) | 5 (5) | 13 (18) | 5 (5) | 5 (11)
VOMITING (Gastrointestinal disorders) | 5 (6) | 7 (8) | 8 (13) | 9 (16) | 12 (16)
ASTHENIA (General disorders) | 3 (3) | 11 (18) | 13 (15) | 6 (11) | 6 (8)
CHEST PAIN (General disorders) | 0 (0) | 7 (9) | 5 (5) | 2 (4) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 15 (19) | 13 (15) | 11 (16) | 10 (10)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
MUCOSAL INFLAMMATION (General disorders) | 1 (3) | 2 (3) | 4 (9) | 5 (6) | 5 (9)
OEDEMA (General disorders) | 1 (1) | 2 (2) | 5 (7) | 0 (0) | 3 (4)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 9 (9) | 9 (12) | 7 (12) | 5 (6)
PAIN (General disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 4 (7) | 8 (13) | 9 (15) | 1 (1) | 9 (12)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
FURUNCLE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IMPETIGO (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (4) | 1 (2) | 4 (8)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (1) | 2 (4) | 4 (5) | 0 (0) | 3 (3)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (4) | 4 (6) | 3 (3) | 4 (5) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 1 (4) | 4 (6) | 3 (4) | 7 (9)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (4) | 3 (5) | 3 (4) | 4 (7) | 6 (7)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (5) | 2 (2) | 3 (5) | 4 (6) | 5 (7)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (2) | 3 (3) | 2 (3) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 6 (6) | 0 (0) | 10 (10) | 5 (11) | 7 (13)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CARBOHYDRATE ANTIGEN 15-3 INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
FIBRIN D DIMER INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
MYOGLOBIN BLOOD INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 2 (2) | 4 (9) | 4 (7)
NEUTROPHIL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
SERUM FERRITIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSFERRIN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 10 (14) | 9 (11) | 4 (4) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (8) | 5 (5) | 3 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 4 (5) | 3 (3)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (9) | 2 (4) | 2 (2) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 6 (6) | 4 (6) | 4 (5)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8) | 6 (8) | 2 (4) | 4 (4)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 4 (5) | 3 (5)
DIZZINESS (Nervous system disorders) | 3 (3) | 8 (9) | 7 (9) | 4 (4) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 4 (4) | 7 (7) | 1 (1) | 2 (3)
DYSMETRIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSTONIC TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (3) | 9 (14) | 7 (14) | 5 (7) | 4 (6)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
HYPOGEUSIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 7 (10) | 4 (4) | 8 (9) | 7 (11)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 5 (9) | 4 (5) | 4 (5) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 9 (12) | 8 (12) | 1 (1) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 3 (3)
INSOMNIA (Psychiatric disorders) | 2 (2) | 7 (8) | 3 (3) | 3 (3) | 4 (5)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
DYSURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 4 (5) | 3 (3) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 2 (3)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (14) | 7 (8) | 6 (7) | 5 (6)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (6) | 7 (12) | 3 (3) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 4 (5) | 7 (8) | 7 (8)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (2) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5) | 19 (20) | 21 (22) | 8 (8) | 10 (10)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 9 (12) | 8 (14) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 6 (7) | 4 (5) | 5 (7)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 3 (4)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 12 (17) | 4 (5) | 4 (9)
RASH (Skin and subcutaneous tissue disorders) | 8 (18) | 5 (6) | 22 (34) | 12 (22) | 17 (22)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (2)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 3 (5) | 4 (7) | 1 (1) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 1 (3) | 4 (4) | 3 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT02322814/Prot_SAP_000.pdf